CLINICAL TRIAL: NCT04518267
Title: Anger and Psychotrauma: Data From Military and Civilians
Acronym: COPMiCiv
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PPRC16; 2020-A00507-32 (Other: IDRCB)
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Civilian group: Participants with civilian status
  Interventions: Behavioral: Structured clinical interview; Behavioral: Psychological questionnaires
- Military group: Participants with military status
  Interventions: Behavioral: Structured clinical interview; Behavioral: Psychological questionnaires

INTERVENTIONS:
Behavioral: Structured clinical interview — A structured clinical interview will be performed at enrollment.
Behavioral: Psychological questionnaires — Several psychological questionnaires will be performed at enrollment.

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) is mainly associated with several emotions such as anger, guilt or shame. By interfering with psychotherapeutic work these emotions can be problematic. When suffering from PTSD, pervasive anger can also have relational consequences. Anger and PTSD are mutually reinforcing: anger can aggravate PTSD symptoms and aggressive behaviours, and conversely, PTSD promotes high levels of anger and aggression. A few explanatory hypotheses have been proposed. In terms of personality factors, anger-treatment may promote the severity of PTSD symptoms and the development of aggressive behaviours. In terms of stressors, exposure to combat and combat-related moral harms could play a role in the relationship between PTSD, anger and traumatic experiences over the course of life. Finally, in clinical terms, in the presence of PTSD, anger and aggressive behaviours may be triggered by substance abuse and depression.

Within the Anglo-Saxon literature, it is recognized that both civilians and military personnel with PTSD exhibit high levels of anger, with a possible predominance among military personnel. While we know that anger management mechanisms can be strongly influenced by cultural aspects and the type of event, there is no data in the French population.

This study proposes to fill in our knowledge of anger-PSTD relationships in the French population and by comparing civilian and military population.

ELIGIBILITY:
Inclusion Criteria:

* To have a PTSD diagnosis
* To be at least 18 years of age

Exclusion Criteria:

* To suffer from trauma-related physical condition (including Traumatic Brain Injury)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of participants suffering from PTSD, half of which will have civilian status and the other half a military status.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Anxiety score | At enrollment
  Spielberger's State-Trait Anger Expression Inventory-II (STAXI-II) will be used to assess anxiety
PTSD severity score | At enrollment
  Clinician-Administered Posttraumatic Stress Disorder Scale (CAPS-5) will be used to assess PTSD severity score. CAPS-5 score may range from 0 to 120 with higher scores meaning greater PTSD severity.
Number of life traumatic events | At enrollment
  Life Event Checklist (LEC) will be used to assess the number of traumatic events experienced by participants throughout their lifetime

SECONDARY OUTCOMES:
Aggressivity score | At enrollment
  Aggressivity Questionnaire (AQ12) will be used to assess aggressivity score. AQ12 score may range from 6 to 72 with higher scores meaning higher aggressivity levels.
Anger Rumination score | At enrollment
  Anger Rumination Scale (ARS) will be used to assess anger rumination score. ARS score may range from 19 to 76 with higher scores corresponding to greater levels of anger rumination.
Alcohol consumption score | At enrollment
  Alcohol Use Identification Test (A.U.D.I.T.) will be used to assess alcohol consumption score Score ≥ 5: at risk use; Score ≥ 8 (7 in women): harmful use; Score ≥ 12 (11 in women): likely alcohol dependence

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Centre hospitalier d'Arras, Arras
  - Centre régional psychotrauma Hauts-de-France, Lille
  - 3ème Centre médical des Armées, Lille
  - Centre Hospitalier de Cadillac, Lormont
  - CHU de Nice, Nice
  - CHU-Lenval hôpitaux, Nice
  - Centre Hospitalier Léon-Jean Grégory de Thuir, Thuir
  - Groupe Hospitalier Paul Guiraud, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided